CLINICAL TRIAL: NCT06159244
Title: Intestinal Microbiota Profiling in HAA Patients
Brief Title: Intestinal Microbiota Profiling in Severe Acute Alcoholic Hepatitis Patients
Acronym: HepathAlc-IM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: CH Montdidier (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2023_843_0123
Record Dates: First submitted 2023-11-21; First posted 2023-12-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Severe Acute Alcoholic Hepatitis; Alcohol; Intestinal Microbiota; Corticosteroids
Keywords: Severe acute alcoholic hepatitis; Alcohol; Intestinal Microbiota; Corticosteroids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- sAH patients (Experimental): the recruitment of patients with sAH will be carried out from the Hepatogastroenterology Service of the University Hospital of Amiens.
  Interventions: Other: stool withdrawal
- Alcohol controls without liver complications (Experimental): the recruitment of alcohol controls will concern patients followed for alcohol addiction without sAH in the antecedents or evolutionary. It will be carried out by the Hospital of Roye-Montdidier. The total number of controls will be equivalent to the number of sAH patients, matched for age and sex.
  Interventions: Other: stool withdrawal
- Healthy non-alcoholic witnesses (Active Comparator): the general population will be called with a matching on age
  Interventions: Other: stool withdrawal

INTERVENTIONS:
Other: stool withdrawal — stool withdrawal at day 0 and day 7

SUMMARY:
In humans, alcohol-related dysbiosis exists with a decrease in bacteroides. This dysbiosis is responsible for the breakdown of the intestinal barrier by a decrease in the synthesis of protective mucus, and some proteins involved in tight junctions or a decrease in defensin (Reg3b, Reg3g) which promotes bacterial growth and ultimately bacterial translocation. The microbiota of a patient with alcoholic hepatitis is different from that of a patient without alcoholic hepatitis. Acute alcoholic hepatitis has a severe prognosis and corticosteroids are the only first line therapy option, with better survival at 28 days versus placebo. However, mortality remains high at 30% at 3 months, which highlights the importance of seeking intestinal microbiota profile on treatment response.

The determination of one or more intestinal microbiota signatures associated with the treatment response Corticosteroids plus FMT or Corticosteroids plus placebo will allow the clinician to have a simple and rapid test obtained in 16S RNA analysis to predict the therapeutic response and potentially the best treatment to adopt and to address medical and medico-economic stakes.

The investigators will first characterize the alcohol-induced dysbiosis by a whole microbiota sequencing in the different groups. Specific bacterial species identify by DNA sequencing should be confirmed by qPCR of 16S rDNA to determine a fingerprint of sAH microbiota. Metabolic properties of intestinal microbiota, such as production of short chain fatty acids, will be analyzed by using HPLC. In the sAH group, evolution of intestinal microbiota will be observed by shotgun DNA sequencing between the day 0 and the day 7 of corticosteroids treatment.

The analysis of sAH patients' microbiota (day 0) will allow us to obtain a non-responder profile to corticosteroids that can be used as a prognostic marker to use in the clinic. The deliverable is the bacterial fingerprint of the treatment response and its valuation is its use as a predictive tool of the response.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 75 years, having :
* Heavy drinker with Maddrey Score ≥ 32 : PT(second)-PT(control)x4.6+Bilirubine (mg/dl)
* Histological confirmed Alcoholic hepatitis
* Personal consent signed to the trial
* No exclusion criteria

Exclusion Criteria:

* Age < 18 years and/or > 75 years,
* Pregnancy or lactating females,
* No personal consent
* Other causes of liver disease: chronic hepatitis B (antigen HBs positive), hepatitis C (HCV RNA positive), acetaminophen hepatotoxicity, biliary obstruction, autoimmune hepatitis, primary biliary cholangitis, primary sclerosis cholangitis, alpha 1 antitrypsine deficiency, and Wilson disease.
* Uncontrolled liver complications:
* Upper gastrointestinal bleed by portal hypertension (4 days required for stable condition)
* Active sepsis (4 days required for stable condition)
* Patient currently treated by antibiotic
* Concomitant Liver cancer (HCC) or extrahepatic malignancy
* Type 1 hepatorenal syndrome (HRS) or renal failure defined as a serum creatinine >221 μmol/L (>2.5 mg/dL) or the requirement for renal replacement therapy
* Grade 4 Hepatic Encephalopathy (HE) by West Haven criteria
* Individuals dependent on inotropic (eg, epinephrine or norepinephrine) or ventilatory support (ie, endotracheal intubation or positive-pressure ventilation)
* Disseminated intravascular coagulation
* Intestinal paralysis
* History of liver transplantation

Other general diseases or severe conditions:

* HIV disease
* Intestinal paralysis
* Intestinal inflammatory disease (Crohn or Ulcerative colitis)
* Clostridium difficilae infection
* Clinical suspicion of pneumonia
* Uncontrolled sepsis
* Acute Alcoholic pancreatitis
* Noncontrolled alcohol withdrawal syndrome
* Cardiac or respiratory bad conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
variation of sample bacterial composition between the three groups | day 7

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No